CLINICAL TRIAL: NCT06866626
Title: The Effect of Harvest Lentil Vegetable Blend Combined with a Theory Based Nutrition Education Intervention on Turkana Children's Health Outcomes
Brief Title: Impact of Harvest Lentil Vegetable Blend and Nutrition Education on Turkana Children's Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: Breedlove Foods Inc (Unknown)
Responsible Party: Principal Investigator, Mary Murimi, Professor of Nutrition, Texas Tech University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB2023-381
Record Dates: First submitted 2025-02-25; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Malnutrition, Child
Keywords: Complementary feeding; WASH practices; Child undernutrition; nutrition education; Harvest Lentil Vegetable Blend; Supplemental feeding
MeSH Terms: conditions — Child Nutrition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): This arm consisted of 171 children aged 6-59 months and 145 children's caregivers. Children received a daily meal of a supplemental food (Harvest Lentil Vegetable Blend) six days a week for a total of eight weeks. Additionally, their caregivers received a theory-based nutrition education intervention on complementary feeding practices and water, hygiene and sanitation (WASH) practices for eight weeks.
  Interventions: Behavioral: Theory-Based Nutrition Education Intervention to Improve Infant and Young Child Feeding Practices and WASH Practices Among Turkana Caregivers; Dietary Supplement: Harvest Lentil Vegetable Blend
- Control group (No Intervention): This group consistent of 147 children aged 6-59 months and 139 children's caregivers. Children in the control group were given one bag of Harvest Lentil Vegetable Blend on the days of data collection while their caregivers received no nutrition education intervention.

INTERVENTIONS:
Behavioral: Theory-Based Nutrition Education Intervention to Improve Infant and Young Child Feeding Practices and WASH Practices Among Turkana Caregivers — This nutrition education intervention was designed following the DESIGN procedure, informed by the Theory of Planned Behavior, and employed health literacy principles. The nutrition education sessions were held Monday through Saturday for a total of 8 weeks in a community building. This nutrition education intervention had 4 modules, module one covered the recommended breastfeeding practices, including early initiation of breastfeeding, exclusive breastfeeding and continued breastfeeding. The second module was on the young child feeding practices, with a focus on the quality and quantity of the child's meal. The third module entailed WASH practices such as disinfection of drinking water, harms of open defecation, and other personal and household hygiene practices. The fourth module served as a comprehensive review of all previous modules.
  Arms: Intervention group
Dietary Supplement: Harvest Lentil Vegetable Blend — Harvest Lentil Vegetable Blend is a dehydrated supplemental food produced from natural ingredients namely, rice, carrots, lentils and onions. This product was prepared by mixing it with water and boiling the mixture for approximately 25-35 minutes to a mid-consistency. In this study we implemented a blanket supplementary feeding program where all the recruited children in the intervention group received a meal of Harvest Lentil Vegetable Blend. The feeding program was on-site, and participating children aged 6-12 months received three-quarters of a cup of the supplemental food, (~ 52 kcal/d). Children aged 13-23 months received 1 cup of the supplemental food (∼69 kcal/d), whereas children aged 24-59 months received 2 cups of the supplemental food (∼138 kcal/d). The feeding was implemented for 6 days a week (Monday through Saturday) for a total of eight weeks.
  Arms: Intervention group

SUMMARY:
The goal of this study was to test the effect of an intervention that Integrated supplemental feeding program for children aged 6-59 months with a caregiver intensive nutrition education intervention on the health outcomes of Turkan children aged 6-59 months.

The purpose of this study was fivefold: (i) to assess child nutrition status, food security status, child feeding practices, water, hygiene and sanitation (WASH) practices, and the associated factors in Turkana County, Kenya. (ii) To assess the nutrition knowledge, attitudes, subjective norms, perceived behavioral control, and intentions towards recommended child feeding practices among Turkana caregivers of children aged 6-59 months. (iii) To assess the effect of a theory-based nutrition education intervention on nutrition knowledge, attitudes, subjective norms, perceived behavioral control, and intentions towards recommended child feeding practices among Turkana caregivers of children aged 6-59 months, (iv) to evaluate the effect of a theory-based nutrition education intervention on child feeding practices and WASH practices among Turkana caregivers of children aged 6-59 months, (v) and to assess the effect of consuming Harvest Lentil Vegetable Blend combined with nutrition education intervention on the nutritional status of Turkana children aged 6 -59 months.

In this quasi-experimental study, children in the intervention group received a daily meal of Harvest Lentil Vegetable Blend (6 days/week) for eight weeks and their caregivers' received sessions of nutrition education on infant and young child feeding practices and WASH practices. The participants in the control group were only given one bag of supplemental food on the days of data collection to compensate for their time

ELIGIBILITY:
Inclusion Criteria:

* Children between 6-59 months
* no known allergy reactions to rice, lentils, carrots and onions
* being a permanent resident of nayada and sopel villages
* willingness to participate in the study

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 602 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Weight | Baseline, midline (4 weeks after baseline assessments) and Endline (8 weeks after baseline assessments)
  Child's weight measurements were taken using an electronic weighing scale (ROTLIN) and recorded to the nearest 0.01kg. To measure the weight of children less than 24 months, we first weighed their caregivers alone and then weighed caregivers with the child. To gain the true weight of the child we subtracted the combined weight of the child and their caregiver from the caregiver's recorded weight. Children older than 24 months were weighed alone.

SECONDARY OUTCOMES:
Height | Baseline, midline (4 weeks after baseline assessments) and Endline (8 weeks after baseline assessments)
  Child's height was measured using Shorr Board® measuring board. For children below 24 months, their lying length was measured. For children older than 24 months, their standing height was taken . Height measurements were recorded to the nearest 0.1cm.
Height-for-age z-scores (HAZ) | Baseline, midline (4 weeks after baseline assessments) and Endline (8 weeks after baseline assessments)
  height-for-age (HAZ) were computed using the WHO Anthro Survey Analyzer software.
Weight-for-age z-scores (WAZ) | Baseline, midline (4 weeks after baseline assessments) and Endline (8 weeks after baseline assessments)
  Weight-for-age z-scores (WAZ) were computed using the WHO Anthro Survey Analyzer software.
Weight-for-height z scores (WHZ) | Baseline, midline (4 weeks after baseline assessments) and Endline (8 weeks after baseline assessments)
  Weight-for-height z-scores (WHZ) were computed using the WHO Anthro Survey Analyzer software.
% of children affected by stunting | Baseline, midline (4 weeks after baseline assessments) and Endline (8 weeks after baseline assessments)
  Children were classified as stunted if their HAZ were below -2 SD the WHO Child Growth Standards
% of children affected by underweight | Baseline, midline (4 weeks after baseline assessments) and Endline (8 weeks after baseline assessments)
  Children were classified as underweight if their WAZ were below -2 SD the WHO Child Growth Standards
% of children affected by wasting | Baseline, midline (4 weeks after baseline assessments) and Endline (8 weeks after baseline assessments)
  Children were classified as wasted if their WHZ were below -2 SD the WHO Child Growth Standards
% of children co-currently affected by wasting and stunting | Baseline, midline (4 weeks after baseline assessments) and Endline (8 weeks after baseline assessments)
  Children were classified as co-currently stunted and wasted if their HAZ and WHZ wew below -2 SD the WHO Child Growth Standards
Meal Frequency | Baseline, midline ( 4 weeks after baseline assessments) and Endline( 8 weeks after baseline assessments)
  The meal frequency was calculated by summing all the feedings a child consumed throughout the day, including solid, semi-solid or soft foods, as well as milk feeds for non-breastfed children. The proportion of children meeting the minimum meal frequency (MMF) was computed among children aged 6-23 months. Per the WHO and UNICEF guidelines, the recommended age-appropriate meal frequency varies both by child's age and breastfeeding status. The recommended MMF is two feedings for breastfed children aged 6-8 months, three feedings for breastfed children 9-23 months, and four feedings for non-breastfed children 6-23 months .
Dietary Diversity | Baseline, midline (4 weeks after baseline assessments) and Endline (8 weeks after baseline assessments)
  To assess children's dietary diversity, caregivers were asked if their children consumed food from the following eight foods groups: (i) breastmilk, (ii) grains, roots, and tubbers (iii) pulses, nuts, and seeds, (iv) dairy products, (v) flesh foods, (vi) eggs, (vii) vitamin-A-rich fruits and vegetables, and (viii) other fruits and vegetables . A food group was assigned a score of one if a child consumed at least one food item from that group; otherwise, it was scored as zero. To calculate the dietary diversity scores, all the food groups consumed were added up. The maximum possible score was eight food groups for children aged 6-23 months and seven food groups for children 24-59 months (excluding breastmilk). A child was considered to have met the minimum dietary diversity if they consumed at least five food groups for ages 6-23 months and at least four food groups for ages 24-59 months .
Consumption of animal sources foods (ASFs) | Baseline, midline (4 weeks after baseline assessments) and Endline (8 weeks after baseline assessments)
  The proportion of children consuming ASFs was calculated by dividing the number of children who consumed at least one food item from dairy products, flesh foods and eggs food groups by the total number of children in the sample.
Acceptable diet score | Baseline, midline ( 4 weeks after baseline assessments) and Endline( 8 weeks after baseline assessments)
  The proportion of children meeting the minimum acceptable diet was calculated among children aged 6-23 months. This is a composite measure of both the dietary diversity and meal frequency . Breastfed children were said to receive minimum acceptable diet if they met both minimum dietary diversity (MDD) and the age-appropriate meal frequency (MMF) . For non-breastfed children they had to meet the MDD, the age-appropriate MMF, and receive at least two milk feeds.
WASH Practices | Baseline, midline ( 4 weeks after baseline assessments) and Endline( 8 weeks after baseline assessments)
  The household WASH practices were assessed using a questionnaire adapted from WHO/UNICEF Joint Monitoring Programme for Water Supply and Sanitation. The assessed WASH practices were: source of drinking water, preparation of drinking water, hand washing at the critical time, proper handwashing technique, sanitation facility and open defecation.
Caregivers' Knowledge on Infant and Child Complementary Feeding Practices | Baseline, midline (4 weeks after baseline assessments) and Endline (8 weeks after baseline assessments)
  A total of 12 items were used to assess caregivers' knowledge on proper IYCF practices. These items have been adapted from the FAO guidelines for assessing nutrition-related knowledge, attitudes, and practices, and were validated by experts in the Community and International Nutrition Research (CINR) Lab. Each correct question was given a score of one, or else a score of zero was given. All the correct scores were summated to provide an aggregate knowledge score for each participant, with the maximum possible score of 12 points. Knowledge scores were further categorized as low (< 6 points), fair (6 - 8 points), and Adequate (> 8 points).
Caregivers' attitudes towards child feeding practices | Baseline, midline (4 weeks after baseline assessments) and Endline (8 weeks after baseline assessments)
  A total of 13 questions were used to assess caregivers' attitudes towards child feeding practices (e.g.: "Solid foods should be introduced to children at 6 months"). Possible responses to the attitudes' questions were "disagree", "not sure", and "agree". The summated attitude scores were calculated for each caregiver, where responses for each question were scored as follows: "disagree" was assigned a score of one, "not sure" a score of two, and "agree" a score of three. The total maximum possible score was 39 points, with a higher score indicating positive attitudes towards child feeding practices . The attitudes scores were further divided into two categories, attitudes towards breastfeeding practices (possible maximum score was 6 points) and attitudes towards complementary practices (possible maximum score was 33 points).
Caregivers perceived social support (subjective norms) | Baseline, midline (4 weeks after baseline assessments) and Endline (8 weeks after baseline assessments)
  Caregivers perceived social support on the practice of proper child feeding practices were assessed using five questions (e.g.: "People who are important to me think that I should start giving my child semisolid or solid foods after he/she turns 2 weeks"). The responses to the subjective norms' questions were on a three-point Likert scale of "disagree", "not sure", and "agree". The aggregate subjective norms score was calculated for each caregiver, where those who responded "disagree" were assigned a score of one, "not sure" assigned a score of two, and "agree" assigned a score of three for positively worded questions and the reverse for the negatively worded questions. The possible maximum subjective norms score was 15 points, and the minimum score was five points. Higher score indicated greater perceived social support for adhering to the recommended child feeding practices.
Caregivers perceived behavioral control | Baseline, midline (4 weeks after baseline assessments) and Endline (8 weeks after baseline assessments)
  Five items were used to assess caregivers perceived behavioral control (e.g.: "I feel confident feeding my child when he/she is sick"). Caregivers answered on three points- Likert scale of "not confident", "ok/so-so", and "confident". The composite perceived behavioral control score was calculated for each caregiver, with those who responded "not confident" assigned a score of one, "ok/so-so" a score of two, and "confident" a score of three. The possible maximum subjective norms score was 15 points and the minimum score was five points, with higher values indicating high perceived behavioral control
Caregivers' intentions to practice recommended child feeding practices | Baseline, midline (4 weeks after baseline assessments) and Endline (8 weeks after baseline assessments)
  A total of five questions were used to assess caregivers' intentions to practice recommended child feeding practices (e.g.: "I intend to feed my child different types of food"). Possible responses to the attitudes' questions were "disagree", "neither agree nor disagree", and "agree". The summative intentions score was calculated for each caregiver, with those who responded "disagree" assigned a score of one, "neither agree nor disagree" a score of two, and "agree" a score of three. The possible maximum subjective norms score was 15 points, with higher values indicating high motivation to comply to the recommended child feeding practices

CONTACTS AND LOCATIONS:
Locations (1):
- Community Building, Sopel Village, Turkana County, Kenya

IPD SHARING:
Plan to Share IPD: No